CLINICAL TRIAL: NCT00341653
Title: A Cohort Study of Smoking Prevention and Health Promotion for Middle School Students in Wuhan, China
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998054; OH98-E-N054
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-05-16

CONDITIONS: Asthma
Keywords: Asthma; Pulmonary Function; Air Pollution; Genetic Polymorphism; Environmental Tobacco Agents
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
We propose to add a collection of buccal cells to a school-based cohort of 7th graders in Wuhan, a large industrial city in China. The cohort study is being conducted by the Wuhan Public Health and Anti-Epidemic Station (Li Yan MD, director and principal investigator). The cohort study is designed to look at several outcomes. One is initiation of smoking. The second is respiratory health in relation to active and passive smoking and other environmental exposures that are prevalent in Wuhan. The respiratory outcomes include changes in pulmonary function, asthma and other respiratory symptoms. Collection of buccal cells is a noninvasive method of obtaining DNA. The addition of a genetic sample will enable us to examine candidate gene associations for asthma and childhood respiratory illness within an interesting and well-characterized Chinese population. In addition, it provides the capability to examine gene environment interaction with respect to common environmental exposures in Wuhan. The ability to examine gene-environment interaction can help to identify relatively subtle effects of pollutants such as environmental tobacco smoke which is becoming a very common exposure due to the major increase in smoking among Chinese men. Other exposures of interest in Wuhan are indoor coal burning and high ambient exposures to particules, ozone and nitrogen oxides. The proposed study has been approved by the human subjects committee of the Wuhan Public Health and Anti-Epidemic Station....

DETAILED DESCRIPTION:
We propose to add a collection of buccal cells to a school-based cohort of 7th graders in Wuhan, a large industrial city in China. The cohort study is being conducted by the Wuhan Public Health and Anti-Epidemic Station (Li Yan MD, director and principal investigator). The cohort study is designed to look at several outcomes. One is initiation of smoking. The second is respiratory health in relation to active and passive smoking and other environmental exposures that are prevalent in Wuhan. The respiratory outcomes include changes in pulmonary function, asthma and other respiratory symptoms. Collection of buccal cells is a noninvasive method of obtaining DNA. The addition of a genetic sample will enable us to examine candidate gene associations for asthma and childhood respiratory illness within an interesting and well-characterized Chinese population. In addition, it provides the capability to examine gene environment interaction with respect to common environmental exposures in Wuhan. The ability to examine gene-environment interaction can help to identify relatively subtle effects of pollutants such as environmental tobacco smoke which is becoming a very common exposure due to the major increase in smoking among Chinese men. Other exposures of interest in Wuhan are indoor coal burning and high ambient exposures to particules, ozone and nitrogen oxides. The proposed study has been approved by the human subjects committee of the Wuhan Public Health and Anti-Epidemic Station.

ELIGIBILITY:
* INCLUSION CRITERIA:

  7th grade students enrolled at the Wuhan Public Health and Anti-Epidemic Station.

Consent signed by parent.

Ages: 12 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5051 (Actual)
Dates: Start 1998-12-01; Study Completion 2019-05-16

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie London, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- Wuhan Public Health and Anti Epidemic Station, Wuhan, China